CLINICAL TRIAL: NCT01754740
Title: The Role of Xerostomia in Burning Mouth Syndrome: Case - Control Study
Acronym: BMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Burning Mouth Syndrome
Keywords: Xerostomia, Salivary flow, Burning Mouth Syndrome.
MeSH Terms: conditions — Burning Mouth Syndrome; Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): 19 patients whom received topical medication of urea 10%
  Interventions: Drug: Uréia
- Control Group (Placebo Comparator): 19 patients whom received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Uréia — The subjects were randomly divided into two groups:
  1. Study Group: 19 patients received topical medication of urea 10% to be applied at the oral cavity 3-4 times per day, during three months.
  Other Names: ureia 10%
  Arms: Study Group
Drug: Placebo — Control Group: 19 patients received placebo (5% sodium carboxymethylcellulose, 0.15% methyl paraben and 10% glycerol in distilled water qsp 100g) to be applied at the oral cavity 3-4 times per day, during three months.
  Arms: Control Group

SUMMARY:
Objectives: to evaluate xerostomia and salivary flow in patients with burning mouth syndrome (BMS) treated with amitriptyline before and after the use of antixerostomic topical medication.

Methods: In this case-control double-blinded study, we enrolled 38 patients with BMS diagnosed according to the (IASP). The subjects were randomly divided into two groups: Study Group: 19 patients whom received topical medication of urea 10% and Control Group: 19 patients whom received placebo to apply at the oral cavity 3-4 times per day, during three months. The patients were evaluated before and after the above treatment. Finally, data were statistically analyzed.

It is know that BMS is eventually associated to reduced salivary flow (Cho et al.,2010; Kho et al., 2010; Marino et al., 2010) and to abnormal salivary composition (increasing concentrations of K+, Na+, Cl-, Ca+2, IgA, amylase) (Patton et al., 2007). Even in the absence of hyposalivation, patients may complain of xerostomia and dry mouth (Cho et al.,2010; Kho et al., 2010; Marino et al., 2010; Thomson, 2005). These patients also have several sensory losses even in taste and smell function, recently described (Siqueira et al., 2006a; Siqueira et al., 2006b; Siviero et al., 2011).

DETAILED DESCRIPTION:
Materials and Methods In this case-control double-blinded study, we enrolled 38 patients with BMS diagnosed according to the International Association for the Study of Pain (IASP) (17), that had been followed at the Craniofacial Pain Clinic of Hospital das Clinicas, School of Medicine of the University of Sao Paulo. All subjects were informed about the purposes of the study, and all signed the informed consent. The protocol had been approved by the local Ethics Committee. No patient had hyposalivation at the moment of diagnosis by the quantitative evaluation. All patients had been treated with 25mg-50mg of amitriptyline within the last three months. They underwent laboratory tests and careful exam to exclude other causes of burning mouth (10).

The exclusion criteria were other facial pain syndromes, other causes for abnormal salivation, other neuropathies or primary diseases associated to burning mouth, inability to answer the questions and / or tests

The subjects were randomly divided into two groups:

1. Study Group: 19 patients received topical medication of urea 10% to be applied at the oral cavity 3-4 times per day, during three months.
2. Control Group: 19 patients received placebo (5% sodium carboxymethylcellulose, 0.15% methyl paraben and 10% glycerol in distilled water qsp 100g) to be applied at the oral cavity 3-4 times per day, during three months.

The patients were evaluated before and after the above treatment with the following instruments:

1. EDOF-HC protocol (Orofacial Pain Clinic - Hospital das Clinicas): a standardized orofacial pain questionnaire to detail: 1) chief complaint, 2) general pain characteristics (location, quality, duration, pain relief, pain triggering), 3) headache and/or body pain complaints, and 4) patient's medical history and co-morbidities (18,19);
2. Xerostomia questionnaire (20);
3. Quantitative sensory testing. All subjects underwent a standardized protocol of quantitative sensory testing (QST) (21) which consists of twelve tests grouped as follows:

   * salivary flow; gustative and olfactory thresholds;
   * thermal detection thresholds for cold and warm sensations;
   * mechanical detection thresholds for touch, vibration and electrical perception;
   * mechanical pain sensitivity including superficial and deep pain thresholds;
   * electric pain threshold at the teeth.
   * corneal reflex.

ELIGIBILITY:
Inclusion Criteria:

* All patients had been treated with 25mg-50mg of amitriptyline within the last three months. They underwent laboratory tests and careful exam to exclude other causes of burning mouth

Exclusion Criteria:

* other facial pain syndromes, other causes for abnormal salivation, other neuropathies or primary diseases associated to burning mouth, inability to answer the questions and / or tests

Ages: 37 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The role of Xerostomia in Burning Mouth Syndrome: case - control study | three years

CONTACTS AND LOCATIONS:
Overall Officials: Silvia RDT Siqueira, Professor, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clinicas, Medical Scholl, University of Sao Paulo, São Paulo, São Paulo, Brazil